CLINICAL TRIAL: NCT00570700
Title: BMS CA180-097: A Phase II Trial of Dasatinib (Sprycel®) in Subjects With Hormone-refractory Prostate Cancer, Previously Treated With Chemotherapy
Brief Title: Trial of Dasatinib (Sprycel®) in Subjects With Hormone-refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Chao Family Comprehensive Cancer Center, Cancer Center, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 06-60; 2007-5564 (Other: University of California, Irvine); BMS CA180-097 (Other: Bristol-Myers Squibb); NCI-2010-00336 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2007-12-06; First posted 2007-12-11 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hormone-refractory Prostate Cancer; Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Prostate Cancer; Recurrent Prostate Cancer
Keywords: prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental): Patients receive oral dasatinib once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 150mg (3 pills) orally daily for as long as the drug benefits
  Other Names: Sprycel®; BMS-354825

SUMMARY:
The purpose of this research study is to find out if a new anti-cancer drug, dasatinib (Sprycel®), previously approved for treatment of some forms of leukemia, will be safe and helpful in treating patients with hormone-refractory prostate cancer.

This is a research study because the study drug, dasatinib (Sprycel®), has not been evaluated for safety or effectiveness in patients with hormone-refractory prostate cancer. The drug is approved by the Food and Drug Administration for treatment of some forms of leukemia; thus, dasatinib (Sprycel®) is not an investigational drug. It has been given safely to hundreds of patients already. However its safety and usefulness in this study population (prostate cancer) is unknown.

Subjects who agree to participate will take 150mg (3 pills) of dasatinib (Sprycel®) daily by mouth for as long as the drug benefits them. During this time, the subject will periodically return to the office for blood/urine tests, X-rays, imaging scans, and/or to complete questionnaires.

DETAILED DESCRIPTION:
Metastatic prostate adenocarcinoma is initially dependent on exogenous androgens for survival and growth; hence, androgen blockade is a key initial intervention for these patients. Whether by orchiectomy or by biochemical blockade, androgen deprivation produces objective regression of prostate cancer in >90% of patients for an average of 1.5-2yrs. Afterwards, however, the remaining prostate cancer cells become independent of exogenous androgen and resume their growth. At this stage the disease is referred to as hormone-refractory prostate cancer (HRPC).

Treatment for HRPC remains unsatisfactory. Only two interventions have been proven through randomized, prospective studies to confer a survival advantage. Docetaxel administered along with prednisone or estramsutine increases overall survival by approximately 3 months, compared with patients treated with mitoxantrone (1,2). In addition, a cell-based vaccine (APC8015) has recently been shown to confer a similar survival advantage for patients with HRPC (3). In 127 patients with HRPC randomized to receive the APC8015 vaccine or unactivated autologous peripheral blood mononuclear cells, there was a 4.5-month increase in median overall survival for the treated cohort (p = 0.01). Thus additional therapeutic tools are needed.

Although the mechanisms whereby androgen-independence develops are not yet fully clarified (7), it is known that malignant progression of prostate cancer involves upregulation of autocrine growth factors and their receptors (8). The process of autocrine reprogramming facilitates autonomous growth and metastasis of the tumor cells. For this reason many of the major novel therapeutic approaches for prostate cancer, currently in clinical trials, are directed against growth factor signaling pathways involving tyrosine kinase receptors and their downstream signaling messengers. Among these, recent evidence suggests a centrol role for the non-receptor tyrosine kinase c-src, in the development, growth, and metastasis of many human cancers (9,10), including prostate carcinomas. Several SFKs are present in prostate cancer cells, including c-src, yes, lck, and lyn (11). SFKs are thought to mediate the signaling pathways of several growth factors and stressors, such as lysophosphatidic acid, bombesin, androgens, and hypoxia (12-15). In prostate cancer cells that are androgen-independent, activation of SFKs is constitutive, rather than ligand-regulated (16). SFKs in turn regulate such diverse prostate cell pathways as VEGF production (15), and FAK signaling (17). Among the response phenotypes mediated by SFKs include cell spreading and attachment, migration and invasion. Genetic and pharmacologic inhibitors of SFKs have been tested on prostate cancer cell lines. Thus two pyrrolopyrimidine c-src inhibitors were shown to inhibit production of the protease MMP-9, as well as the functional ability of the cells to invade Matrigel (18). These phenotypes occurred at inhibitor concentrations that did not significantly affect cell proliferation. In contrast a peptide inhibitor of the lyn kinase inhibited the proliferation of prostate cancer cell lines in culture, and reduced the growth of DU145 xenografts in nude mice (19). Thus a spectrum of responses have been seen in prostate cancer cells or tumors treated with SFK inhibitors, including inhibition of growth.

ELIGIBILITY:
Inclusion Criteria:

* Must have biopsy-proven adenocarcinoma of the prostate
* Must have hormone-refractory prostate cancer, defined as an increasing PSA by >= 3 ng/ml from androgen-blockade nadir, or new measurable or evaluable lesion on imaging studies, after treatment with orchiectomy, luteinizing hormone-releasing hormone (LHRH) agonist, antiandrogen or diethylstilbestrol (DES)
* Subjects must have received at least one cycle of single-agent or combination chemotherapy for hormone refractory prostate cancer (HRPC), last administered at least 4 weeks prior to the start of dasatinib
* Subjects may not have received more than one type (single agent or combination) of chemotherapy regimen; subjects may include (but are not limited to) the following: HRPC subjects who were treated with palliative chemotherapy and either failed to respond, or responded for a period of time but now have worsening disease (i.e. relapsed/refractory to chemotherapy); HRPC subjects who were treated with palliative chemotherapy but stopped treatment because of toxicity (i.e. intolerant of chemotherapy); HRPC subjects who have been treated with palliative chemotherapy with response, whose chemotherapy has been interrupted, and who now have evidence of progressive disease (i.e. potentially chemotherapy responsive but subject does not desire to restart cytotoxic drugs)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of at least 8 weeks, based on clinical judgment of the treating physician
* Adequate hematologic, renal and liver function as evidenced by the following (subjects may have lower hematologic parameters if the cytopenias are thought by the treating physician to be secondary to marrow involvement by prostate cancer):
* white blood cell count (WBC) > 2.0 bil/L; grade 0-1
* absolute neutrophil count (ANC) > 1.0 bil/L; grade 0-1
* Platelets > 100 bil/L; grade 0-1
* Hemoglobin > 8.0gm/dL
* Creatinine < 1.5x upper limit of normal (ULN)
* Prothrombin time (PT), Partial Thromboplastin Time (PTT) < 1.2 x ULN; grade 0-1
* Total bilirubin < 2x ULN
* aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 2.5x ULN
* Na, K, Mg, P, Ca >= lower limit of normal
* Elevated PSA level (at least 3 ng/mL), or measurable prostate cancer by CT or MRI scans (PSA level must have shown two consecutive increases [at >= 14 day intervals] since the previous nadir)
* Ability to take oral medication (dasatinib must be swallowed whole)
* Subjects of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped
* Signed informed consent documents including Health Insurance Portability and Accountability Act (HIPAA) according to institutional guidelines
* Concomitant Medications: Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (in addition Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia)

Exclusion Criteria:

* Subjects should have had no chemotherapy within 4 weeks of the start of treatment with dasatinib
* Prior localized radiotherapy for metastatic disease is permitted, provided the treatment volume is less than25% of potential marrow space (the radiotherapy must have been completed 6 weeks prior to enrollment)
* Systemic radiotherapy with samarium-153 must have been completed at least 2 months prior to enrollment (subjects may not have received prior strontium-89 [Metastron] therapy)
* At least 6 weeks have elapsed from the last dose of cytotoxic or targeted therapeutics to the time of prescreening; if the subject has received a combination regimen of standard chemotherapy plus an investigational agent, a 6 week washout period is required
* Subjects may not have received treatment with any kinase inhibitor
* At least 2 months must have elapsed from time of dosing with vaccines to the time of prescreening
* No malignancy, other than prostate cancer, that required radiotherapy or systemic treatment within the past 5 years
* Subjects may not have any of the following: Clinical evidence of uncontrolled heart failure, myocardial infarction, or angina within the previous 6 months; prolonged QT interval Fridericia's (QTcF) > 450msec; history of unstable ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation, or torsades de pointes); concomitant use of drugs known to cause torsades de pointes [quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycins, clarithromycin, chlorpromazine, haloperidol, mesoridazine,thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine] (these agents must have been discontinued at least 7 days prior to starting dasatinib); subjects with hypokalemia or hypomagnesemia are excluded if the electrolyte anomaly cannot be corrected
* Subjects may not be enrolled with any of the following: History of a significant bleeding disorder unrelated to cancer, including diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), and diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies); GI bleeding from any cause within 3 months; Concomitant use of anticoagulants, except for low-dose warfarin (for prophylaxis to prevent catheter thrombosis) or heparin flushes (for IV lines), is prohibited (Note that chronic use of aspirin is prohibited)
* Subjects must meet the following restrictions: Subjects may not have a concurrent medical condition which may increase the risk of toxicity, including pleural or pericardial effusion of any grade, or uncontrolled hypertension; Concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended (The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy); Patient must discontinue St. Johns Wort while receiving dasatinib therapy; Subjects must not use intravenous bisphosphonates during the first 8 weeks of dasatinib therapy due to risk of hypocalcemia; Subjects may not be receiving any restricted cytochrome P450 3A4 (CYP3A4) inhibitors (If the investigator feels that any of these agents should be given as uniquely useful for a clear diagnosis, the situation should be discussed with the Principal Investigator, and a clear monitoring program should be planned)
* Subjects may not have evidence of untreated intracranial metastases, or untreated prostate cancer producing spinal cord compression

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Lilly, MD, FACP, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (6):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - St. Joseph Hospital, Orange, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, and Hollings Cancer Network, Charleston, South Carolina

REFERENCES:
- [Result] Twardowski PW, Beumer JH, Chen CS, Kraft AS, Chatta GS, Mitsuhashi M, Ye W, Christner SM, Lilly MB. A phase II trial of dasatinib in patients with metastatic castration-resistant prostate cancer treated previously with chemotherapy. Anticancer Drugs. 2013 Aug;24(7):743-53. doi: 10.1097/CAD.0b013e328361feb0. PMID 23652277

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dasatinib
Started | 38
Completed | 27
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 68 [55 to 88]
Sex/Gender, Customized [Number; unit: participants]
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 26
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Disease Control (DC) (Based on PSA, Bone Scan, FACT-P, RECIST)
Description: A "positive effect" will be defined as a complete response, partial response, or stable disease. "Lack of positive effect" will be defined as progressive disease. Subjects with a mixed response should be continued on therapy until they either fulfill the criteria for positive effect or lack of positive effect, with evaluation every 56 days.
  The disease control (DC) rate was evaluated as a composite endpoint of the treatment effect on four parameters: 1) Prostate-specific antigen (PSA), 2) measurable disease (if present) by RECIST criteria, 3) bone scan, and 4) quality-of-life as measured by the FACT-P questionnaire.
Time Frame: From day 56 (8 weeks) and every 8 weeks thereafter until the date of first documented progression or date of death from any cause, whichever came first, assessed until death, the patient withdraws consent, or the study ends, up to 2 years
Population: 27 subjects were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 27
Participants | 5

2. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression, defined as the interval from the first day of dasatinib treatment until either (1) there has been a 50% increase in PSA above the treatment nadir, with a minimum of 5ng/mL, or (2) a 25% increase in PSA level above pretreatment levels, with a minimum of 5ng/mL. All PSA-based assessments require a confirmatory level no more than 1 month later.
Time Frame: From initial date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
Population: Data not collected due to relatively poor drug tolerance and relatively rapid PSA increases in most patients as it was not feasible to continue patients on treatment.
Arm/Group | Dasatinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Subjects With Dasatinib Toxicity Using Common Terminology Criteria (CTC) (v. 3.0)
Description: Due to relatively poor drug tolerance and relatively rapid PSA increases in most patients it was not feasible to continue patients on treatment until there was radiographic evidence of disease progression.
Time Frame: From initial date of treatment through study completion, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 27
Participants | 12

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Dasatinib
All-Cause Mortality (participants affected / at risk) | 8/38
Serious Adverse Events (participants affected / at risk) | 17/38
Other Adverse Events (participants affected / at risk) | 11/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=38)
Fatigue/asthenia (General disorders) | 5 — Grade 3 Fatigue/asthenia in 5 (19%) of subjects.
Diarrhea (Gastrointestinal disorders) | 2 — Grade 3 Diarrhea occurred in 2 (8%) of subjects.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 — Grade 3 Dyspnea occurred in 2 (8%) subjects.
GI bleed (Gastrointestinal disorders) | 2 — Grade 3 GI bleed occurred in 2 (8%) subjects.
Hyponatremia (Blood and lymphatic system disorders) | 2 — 1 (4%) Grade 3 and 1 (4%) Grade 4 Hyponatremia event occurred.
Elevated lipase (Blood and lymphatic system disorders) | 1 — Grade 3 Elevated lipase occurred in 1 (4) subject.
Pleural / pericardial effusion (Cardiac disorders) | 1 — Grade 3 Pleural / pericardial effusion occurred in 1 (4%) subject.
Anemia (Blood and lymphatic system disorders) | 1 — Grade 3 Anemia occurred in 1 (4%) subject.
Venous thrombosis (Blood and lymphatic system disorders) | 1 — Grade 3 Venous thrombosis occurred in 1 (4%) subject.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=38)
Anorexia (Psychiatric disorders) | 2
Decreased Appetite (Psychiatric disorders) | 3
Elevated Alkaline Phosphatase Levels (Blood and lymphatic system disorders) | 3
Elevated Amylase (Blood and lymphatic system disorders) | 4
Elevated Aspartate Aminotransferase Levels (Blood and lymphatic system disorders) | 3
Elevated lipase levels (Blood and lymphatic system disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 3
Fatigue (General disorders) | 6
Diarrhea (Gastrointestinal disorders) | 3
Nausea (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Headache (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes